CLINICAL TRIAL: NCT03963037
Title: Characterization of Two Novel Truncating Mutations in the Apob Gene Leading to Hypobetalipoproteinemia: A Pilot Study
Brief Title: Characterization of Two Novel Mutations in the Apob Gene
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 20190130-1943
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Familial Hypobetalipoproteinaemia - Heterozygous Form; Low-LDL-syndrome
Keywords: Apolipoprotein B; Cholesterol; Lipoprotein; Metabolism; Steatosis; Cirrhosis; Hepatocellular Carcinoma
MeSH Terms: conditions — Fatty Liver; Fibrosis; Carcinoma, Hepatocellular | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: The family members of our two kindreds who carry the truncating mutation in the Apolipoprotein B gene.
  Interventions: Other: Blood draw
- Controls: The family members of our two kindreds who are no carriers of the truncating mutation in the Apolipoprotein B gene.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Draw venous blood for baseline blood parameters and plasma samples for lipoprotein fractionation.

SUMMARY:
The pilot study has the target to evaluate the outcomes of two novel mutations in the gene of Apolipoprotein B (ApoB). ApoB is the main part of the low-density lipoprotein (LDL). LDL is the main transporter of cholesterol from the liver to the periphery. The two novel mutations lead to a heavily truncated Apolipoprotein B. Therefore the patients show severely decreased ApoB and LDL-Cholesterol levels. The acquired disease is known as "Familial Hypobetalipoproteinemia". Beside the protection from cardiovascular disease due to decreased LDL-Cholesterol, patients tend to show elevated serum aminotransferases, fatty liver and occasional cases of cirrhosis and carcinoma.

To elucidate the differences in lipoprotein assembly the investigators aim to characterize the changes due to the mutations in the patients. Family members not carrying the mutations are the control group. The assessment includes lipoprotein fractionation, MRI scans of the liver and a thorough assessment of medical history of all patients to look for potential side effects of the mutation.

The only intervention needed for the study is to draw blood samples of every participant. The necessary positive vote from the ethics committee of the Medical University of Innsbruck is given.

ELIGIBILITY:
Inclusion Criteria:

* Full legal age
* Written Informed Consent
* Diagnosed hypobetalipoproteinemia
* Exception of it are the controls
* Controls have to be family members
* Exclusion of a truncating mutation in the ApoB gene

Exclusion Criteria:

* No diagnosed hypobetalipoproteinemia
* No truncating mutation in the Apo B gene
* Exception of it ar the controls

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants descend from two families. Each family carries a novel truncating mutation in the ApoB gene. The family members decided to participate in our pilotstudy to elucidate the changes caused by the mutations. Familial hypobetalipoproteinemia is a codominant disorder, so family members not carrying the mutations serve as control group.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Difference in lipoprotein profiles | 6 months
  Lipoprotein profiles are measured via Fast Protein Liquid Chromatography in both groups and compared.
Differences in amounts of liver fat | 12 months
  Liver fat is non-invasive quantified by MRI scan
Differences in HDL-efflux | 6 months
  Compare the results between groups of HDL-efflux assays

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Ebenbichler, MD, Prof., Principal Investigator — Department of Internal Medicine I, Medical University of Innsbruck, Austria
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

REFERENCES:
- [Background] Welty FK. Hypobetalipoproteinemia and abetalipoproteinemia. Curr Opin Lipidol. 2014 Jun;25(3):161-8. doi: 10.1097/MOL.0000000000000072. PMID 24751931
- [Background] Di Costanzo A, Di Leo E, Noto D, Cefalu AB, Minicocci I, Polito L, D'Erasmo L, Cantisani V, Spina R, Tarugi P, Averna M, Arca M. Clinical and biochemical characteristics of individuals with low cholesterol syndromes: A comparison between familial hypobetalipoproteinemia and familial combined hypolipidemia. J Clin Lipidol. 2017 Sep-Oct;11(5):1234-1242. doi: 10.1016/j.jacl.2017.06.013. Epub 2017 Jun 24. PMID 28733173
- [Background] Schonfeld G. Familial hypobetalipoproteinemia: a review. J Lipid Res. 2003 May;44(5):878-83. doi: 10.1194/jlr.R300002-JLR200. Epub 2003 Mar 16. PMID 12639976
- [Background] Hooper AJ, Heeks L, Robertson K, Champain D, Hua J, Song S, Parhofer KG, Barrett PH, van Bockxmeer FM, Burnett JR. Lipoprotein Metabolism in APOB L343V Familial Hypobetalipoproteinemia. J Clin Endocrinol Metab. 2015 Nov;100(11):E1484-90. doi: 10.1210/jc.2015-2731. Epub 2015 Aug 31. PMID 26323024